CLINICAL TRIAL: NCT05211908
Title: Clinical Performance of Different Adhesive Strategies With a Universal System in Sclerosed Dentin in NCCL: A Double-blind Randomized Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Clinical professor, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara-0013
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Sclerotic Dentine; Non Carious Cervical Lesion
Keywords: adhesives; dental bonding
MeSH Terms: conditions — Dentin, Secondary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- D-SE (Experimental): Absence of dentinal sclerosis and self-etching adhesive protocol
  Interventions: Procedure: Composite resin restoration with Self Etch adhesive protocol and absence of sclerotic dentin
- D-SELETIVE (Active Comparator): Absence of dentinal sclerosis and selective enamel etching adhesive protocol
  Interventions: Procedure: Composite resin restoration with Seletive enamel etch adhesive protocol and absence of sclerotic dentin
- SD-SE (Experimental): Sclerotic dentin and self-etching adhesive protocol
  Interventions: Procedure: Composite resin restoration with Self Etch adhesive protocol and presence of sclerotic dentin
- SD-SELETIVE (Experimental): Sclerotic dentin and selective enamel etching adhesive protocol
  Interventions: Procedure: Composite resin restoration with Seletive enamel etch adhesive protocol and presence of sclerotic dentin

INTERVENTIONS:
Procedure: Composite resin restoration with Self Etch adhesive protocol and absence of sclerotic dentin — The adhesive system Single Bond Universal (3M Oral Care; Brazil) and a nanoparticulate composite resin Z350 XT (3M Oral Care; Brazil), shade A3B, will be the materials used in the restorative procedures.
  For the D-SE group, the universal adhesive system will be applied with a disposable microbrush, actively, for 20s and then a gentle stream of air will be used for 5s to solvent evaporation, followed by light curing for 10s using the Valo Cordless light curing (Ultradent Products Inc.), in Standard mode (1000mW /cm2).
  All groups will receive the restorations made following the incremental technique of insertion of composite resin (2mm per increment), which will be light cured according to the manufacturer's recommendations.
  Arms: D-SE
Procedure: Composite resin restoration with Seletive enamel etch adhesive protocol and absence of sclerotic dentin — The adhesive system Single Bond Universal (3M Oral Care; Brazil) and a nanoparticulate composite resin Z350 XT (3M Oral Care; Brazil), shade A3B, will be the materials used in the restorative procedures.
  For the D-SELETIVE group a 37% phosphoric acid will be applied only at the enamel margin for 15s, then rinsed with water for 20s, and slightly dry. The universal adhesive system will be applied with a disposable microbrush, actively, for 20s and then a gentle stream of air will be used for 5s to solvent evaporation, followed by light curing for 10s using the Valo Cordless light curing (Ultradent Products Inc.), in Standard mode (1000mW /cm2).
  All groups will receive the restorations made following the incremental technique of insertion of composite resin (2mm per increment), which will be light cured according to the manufacturer's recommendations.
  Arms: D-SELETIVE
Procedure: Composite resin restoration with Self Etch adhesive protocol and presence of sclerotic dentin — The adhesive system Single Bond Universal (3M Oral Care; Brazil) and a nanoparticulate composite resin Z350 XT (3M Oral Care; Brazil), shade A3B, will be the materials used in the restorative procedures.
  For the SD-SE group, the universal adhesive system will be applied with a disposable microbrush, actively, for 20s and then a gentle stream of air will be used for 5s to solvent evaporation, followed by light curing for 10s using the Valo Cordless light curing (Ultradent Products Inc.), in Standard mode (1000mW /cm2).
  All groups will receive the restorations made following the incremental technique of insertion of composite resin (2mm per increment), which will be light cured according to the manufacturer's recommendations.
  Arms: SD-SE
Procedure: Composite resin restoration with Seletive enamel etch adhesive protocol and presence of sclerotic dentin — The adhesive system Single Bond Universal (3M Oral Care; Brazil) and a nanoparticulate composite resin Z350 XT (3M Oral Care; Brazil), shade A3B, will be the materials used in the restorative procedures.
  For the SD-SELETIVE group a 37% phosphoric acid will be applied only at the enamel margin for 15s, then rinsed with water for 20s, and slightly dry. The universal adhesive system will be applied with a disposable microbrush, actively, for 20s and then a gentle stream of air will be used for 5s to solvent evaporation, followed by light curing for 10s using the Valo Cordless light curing (Ultradent Products Inc.), in Standard mode (1000mW /cm2).
  All groups will receive the restorations made following the incremental technique of insertion of composite resin (2mm per increment), which will be light cured according to the manufacturer's recommendations.
  Arms: SD-SELETIVE

SUMMARY:
The aim of this randomized, prospective, parallel, double-blind clinical trial will be to evaluate the clinical performance of restorations performed in non-carious cervical lesions (NCCL) using a soft ph universal adhesive system, varying the adhesive strategy (self-etching vs. selective etching of the enamel) and the sclerosis characteristics of the dentinal substrate over 24 months.

DETAILED DESCRIPTION:
Two hundred restorations will be performed in NCCL of volunteers of both genders, by a single operator, using the Single Bond Universal(3M ESPE) adhesive system. The restorations will be randomly allocated into 4 groups (n-50): D-SE (absence of dentinal sclerosis and self-etching protocol); D-SELETIVE (absence of dentinal sclerosis and selective enamel etching protocol); SD-SE (sclerotic dentin and self-etching protocol); SD-SELETIVE (sclerotic dentin and selective enamel etching protocol). The randomization process within subject was performed by computer-generated tables by a staff member not involved in the research protocol. Details of the allocated group were recorded on cards contained in sequentially numbered, opaque, sealed envelopes. These were prepared by a staff member who was not involved in any of the phases of the clinical trial. The allocation assignment was revealed by opening the envelope on the day of the restorative procedure.The operator was not blinded to group assignment when administering.

The evaluations of the clinical performance of the restorations will be carried out by two previously calibrated examiners, adopting the criteria of the United States Public Health Service (USPHS) for the variables retention, marginal adaptation, marginal staining and postoperative sensitivity . The intragroup statistical analysis will be performed using the McNemar test for the variables retention and postoperative sensitivity; and by Wilcoxon for adaptation and marginal staining. To compare the clinical performance inter groups in the different assessment intervals, Fisher's exact test (retention and postoperative sensitivity) and Kruskal-Wallis (adaptation and marginal staining) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Good general health status
* Good oral hygiene
* Absence of periodontal disease
* Minimum of 20 teeth in occlusion
* Presence at least one (01) non-carious cervical lesion in a tooth with pulp vitality.
* Non-carious cervical lesion greater than 1mm in depth.
* Non-carious cervical lesion involving enamel and dentin.

Exclusion Criteria:

* Non- carious cervical lesion cavo surface margin involving more than 50% of the enamel.
* NCCL in crack teeth.
* Absence of opposing teeth and/or adjacent to the lesion.
* Presence of occlusal trauma in the NCCL tooth
* Presence of orthodontic appliance or removable partial denture with retention in the tooth where the lesion is located
* Patients that underwent tooth whitening procedures within a period of less than 14 days from the date of restoration
* Patients with high risk of caries (presence of three or more active caries lesions)
* Xerostomia
* Bruxism
* Pregnant women
* Patients who do not accept the study conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Retention | 1 year
  The restorations retention will be evaluated according to the criteria established by the United States Public Health Service (USPHS), classifying them in the following scores:
  Alpha - retained Bravo - partially retained Charlie - restoration lost For evaluation of clinical performance, beta and charlie scores will be considered as failure.
Retention | 2 years
  The restorations retention will be evaluated according to the criteria established by the United States Public Health Service (USPHS), classifying them in the following scores:
  Alpha - retained Bravo - partially retained Charlie - restoration lost For evaluation of clinical performance, beta and charlie scores will be considered as failure.

SECONDARY OUTCOMES:
Marginal adaptation | 1 year
  Marginal adaptation will be evaluated according to the criteria established by the United States Public Health Service (USPHS), classifying them in the following scores:
  Alpha - Restoration is continuous with existing anatomic form. Bravo - Detectable V-shaped defect in enamel only. Catches explorer going both ways Charlie - Detectable V-shaped defect to dentin-enamel junction
Marginal adaptation | 2 years
  Marginal adaptation will be evaluated according to the criteria established by the United States Public Health Service (USPHS), classifying them in the following scores:
  Alpha - Restoration is continuous with existing anatomic form. Bravo - Detectable V-shaped defect in enamel only. Catches explorer going both ways Charlie - Detectable V-shaped defect to dentin-enamel junction
Marginal staining | 1 Year
  Marginal staining will be evaluated according to the criteria established by the United States Public Health Service (USPHS), classifying them in the following scores:
  Alpha - No discoloration along the margin Bravo - Slight and superficial staining (removable, usually localized). Charlie - Deep staining cannot be polished away
Marginal staining | 2 Years
  Marginal staining will be evaluated according to the criteria established by the United States Public Health Service (USPHS), classifying them in the following scores:
  Alpha - No discoloration along the margin Bravo - Slight and superficial staining (removable, usually localized). Charlie - Deep staining cannot be polished away

CONTACTS AND LOCATIONS:
Overall Officials: Cecy M Silva, PhD, Principal Investigator — Universidade Federal do Pará
Locations (1):
- Universidade Federal do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No